CLINICAL TRIAL: NCT03998046
Title: Coordinating Pragmatic Primary Care Population Management for Obesity
Acronym: C3PO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ronald Ackermann, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STU00207153; R34DK114773 (NIH)
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Results first posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-01

CONDITIONS: Obesity; Cardiovascular Risk Factor
Keywords: overweight; obesity; prediabetes; type 2 diabetes; hypertension; dyslipidemia; cardiovascular risk factor; adult; primary care
MeSH Terms: conditions — Obesity; Overweight; Prediabetic State; Diabetes Mellitus, Type 2; Hypertension; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: The active intervention "C3PO" involves enhanced use of pragmatic electronic health record system technologies and members of the primary care workforce to increase supportive accountability and problem solving support for weight loss goals and behavior, which in turn will lead to routine self-weighing, increased take up into intensive community programs, and increased adoption and maintenance of healthy eating and physical activity behaviors that collectively lead to greater weight loss at a population level.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients will be randomized to either Basic Resources and Services or the C3PO intervention arm. Although patients will be aware of the specific forms of support they are receiving throughout the trial, each individual will not be aware that they are part of a randomized experiment and will not know that other patients may be receiving different levels of support. For this reason, the non-concealed nature of the behavioral support intervention for participating patients should not introduce bias. Investigators and outcome assessors will not be aware of intervention assignment during the study conduct or evaluation phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic Resources and Services (Active Comparator): Patients will receive outreach engagement in goal setting via MyChart, an electronic scale, telemonitoring of self weighing, and information about linkages to extant intensive lifestyle interventions in the community
  Interventions: Behavioral: Outreach Support for Weight Loss Goal Setting and Self-Weighing; Behavioral: Outreach Decision Support to Encourage Linkages to Intensive Community Lifestyle Interventions
- Coordinated Primary Care Population Management (C3PO) (Experimental): Patients will receive outreach engagement in goal setting via MyChart, an electronic scale, telemonitoring of self weighing, information about linkages to extant intensive lifestyle interventions, and outreach MyChart messages that are tailored to each individual's pattern of self-weighing and progress towards their weight goal, and more intensive support from a primary care nurse based on self-weighing behavior and weight loss success.
  Interventions: Behavioral: Outreach Support for Weight Loss Goal Setting and Self-Weighing; Behavioral: Outreach Decision Support to Encourage Linkages to Intensive Community Lifestyle Interventions; Behavioral: Adaptive Tailoring of Information Delivery and Intensity of Primary Care Outreach Support

INTERVENTIONS:
Behavioral: Outreach Support for Weight Loss Goal Setting and Self-Weighing — Patients will receive a MyChart activation message assessing weight loss interest that invites them to complete a MyChart Survey encouraging a weight loss goal using principles adapted from Brief Action Planning. Patients will then receive a cellular network-enabled electronic body weight scale, and weighing data transmitted by the scale will be received and integrated into the electronic health record for access by the patient's primary care team.
Behavioral: Outreach Decision Support to Encourage Linkages to Intensive Community Lifestyle Interventions — Patients will receive via MyChart information and decision support designed to encourage linkages to and participation in intensive lifestyle programs available in the community. Patients who request information or clinical referrals will also receive them. "Refreshes" of community linkage information will be sent by MyChart every 1 to 4 weeks.
Behavioral: Adaptive Tailoring of Information Delivery and Intensity of Primary Care Outreach Support — Data received into the electronic health record from the cellular network-enabled electronic scale will categorize each patient based on their daily self-weighing behaviors and rate of progress towards their weight loss goal. Patients who are not engaged in daily self-weighing or are not making progress towards their goal will receive more intensive outreach support in the form of automated weekly MyChart problem solving messages, more frequent encouragement to access a broader array of community resources, and telephonic support from a nurse care coordinator who is an existing member of the primary care team. Support from this nurse care coordinator will be facilitated by the incorporation of each patient's self-weighing data into an EpicCare patient dashboard accessible to the nurse coordinator and other members of the care team
  Arms: Coordinated Primary Care Population Management (C3PO)

SUMMARY:
The C3PO pilot and feasibility study uses a rigorous, mixed-method research design to provide information needed to refine and implement a technology-mediated primary care outreach intervention approach before conducting a larger and more definitive future intervention trial.

DETAILED DESCRIPTION:
This study will implement and evaluate a pragmatic and generalizable framework for population management of obesity by the primary care sector. With patient and other stakeholder input, the C3PO intervention will be designed to leverage existing primary care professionals and technologies to implement a scalable framework for population obesity management that coordinates primary care services with extant intensive lifestyle interventions in community settings to achieve wider reach and population-level effectiveness. A rigorous, mixed-method pilot and feasibility study will provide critical information needed to optimize the intervention design and prepare us for a larger and definitive future trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27 kg/m2
* ≥ 1 CVD risk condition (hypertension, dyslipidemia, prediabetes or type 2 diabetes)
* Registered in Northwestern Medical Group's EpicCare MyChart patient portal
* Received and completed MyChart survey of weight loss interest
* Affirms interest in weight loss goal setting and receiving additional resource information and electronic Scale.

Exclusion Criteria:

* Evidence of hospitalization in past 30 days
* Most recent blood pressure >180/105
* Cancer (non-skin) treatment within the past 2 years
* Encounter diagnosis for hypoglycemia in past 30 days
* Actively receiving care from the bariatric surgery service or a bariatric medication order in the past 100 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Basic Resources and Services: Patients received outreach engagement in goal setting via MyChart, an electronic scale, telemonitoring of self weighing, and information about linkages to extant intensive lifestyle interventions in the community
- Coordinated Primary Care Population Management (C3PO): Patients received outreach engagement in goal setting via MyChart, an electronic scale, telemonitoring of self weighing, information about linkages to extant intensive lifestyle interventions, and outreach MyChart messages that are tailored to each individual's pattern of self-weighing and progress towards their weight goal, and more intensive support from a primary care nurse based on self-weighing behavior and weight loss success.
Period: Overall Study
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO)
Started | 38 | 42
Completed | 38 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO) | Total
Number analyzed (Participants) | 38 | 42 | 80
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 8 | 4 | 12
  45-64 years | 18 | 26 | 44
  65+ years | 12 | 12 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 12 | 18 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 3 | 8 | 11
  Black | 12 | 11 | 23
  Asian | 2 | 4 | 6
  White | 16 | 18 | 34
  Other | 5 | 1 | 6
Pre-diabetes [Count of Participants; unit: Participants] — Number of patients with a pre-diabetes diagnosis in clinical record
  Participants | 19 | 11 | 30
Diabetes [Count of Participants; unit: Participants] — Type-2 Diabetes Mellitus diagnosis and/or recent diabetes class medication order in clinical record.
  Participants | 6 | 13 | 19
High blood pressure [Count of Participants; unit: Participants] — Hypertension diagnosis and/or recent anti-hypertensive medication order in clinical record.
  Participants | 29 | 33 | 62
Hyperlipidemia [Count of Participants; unit: Participants] — Diagnosis of hyperlipidemia and/or recent anti-lipidemic class medication in medical record.
  Participants | 27 | 34 | 61
Baseline clinical weight [Mean (Standard Deviation); unit: lbs.] | 209.2 (40.5) | 205.9 (35.6) | 207.5 (37.8)
Hemoglobin A1C [Mean (Standard Deviation); unit: Percent of HbA1C] — Population: Clinical A1c values were not available for all participants
  Percent of HbA1C
    number analyzed (Participants) | 33 | 34 | 67
    (all) | 6.03 (0.90) | 6.29 (1.35) | 6.16 (1.15)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 136.89 (18.25) | 132.83 (17.72) | 134.76 (17.98)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Population: Clinical total cholesterol values were not available for all participants.
  mg/dL
    number analyzed (Participants) | 37 | 41 | 78
    (all) | 183.22 (41.04) | 187.27 (49.21) | 185.35 (45.27)
Non-HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Population: Clinical Non-HDL Cholesterol values not available for all participants.
  mg/dL
    number analyzed (Participants) | 37 | 41 | 78
    (all) | 127.08 (35.23) | 133.46 (45.56) | 130.44 (40.85)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved 5% Weight Loss Goal at 6 Months
Description: Proportion of Participants who Reach a 5% Weight Loss Goal at 6 Months, calculated as the percent of all participants for whom the following calculation is greater than or equal to 5%: (Baseline body mass (kg) - Body mass measured at 6 months (kg))/(Baseline body mass (kg))
Time Frame: Baseline - 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO)
Number analyzed (Participants) | 38 | 42
Participants | 6 | 6
Statistical Analysis 1: Comparison: Basic Resources and Services vs Coordinated Primary Care Population Management (C3PO); Test type: Superiority; p = .85, Chi-squared

2. Secondary Outcome: Costs to Implement the Intervention
Description: Costs (US$) of Intervention Components, including the costs to fund personnel efforts, technology, and other intervention components
Time Frame: Baseline - 12 Months
Population: Intervention cost inputs include personnel, supplies, contract services, and facility and administrative costs, all from the perspective of the health system. Research-only costs were excluded from intervention cost estimations.
Measure: Number; unit: US Dollars per enrolled participant
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO)
Number analyzed (Participants) | 38 | 42
US Dollars per enrolled participant | 423 | 572

3. Secondary Outcome: Change in Hemoglobin A1C
Description: Mean change in Hemoglobin A1C levels (DCCT%) from baseline to 12 months
Time Frame: Baseline - 12 Months
Measure: Mean (Standard Deviation); unit: Percent of HbA1C
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO)
Number analyzed (Participants) | 33 | 34
Percent of HbA1C | -.11 (.42) | .09 (.80)
Statistical Analysis 1: Comparison: Basic Resources and Services vs Coordinated Primary Care Population Management (C3PO); Test type: Superiority; p = .20, t-test, 2 sided

4. Secondary Outcome: Change in Systolic Blood Pressure
Description: Mean change in systolic blood pressure (mmHg) from baseline to 12 months
Time Frame: Baseline - 12 Months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO)
Number analyzed (Participants) | 38 | 42
mmHg | -3.34 (18.09) | .45 (20.06)
Statistical Analysis 1: Comparison: Basic Resources and Services vs Coordinated Primary Care Population Management (C3PO); Test type: Superiority; p = .38, t-test, 2 sided

5. Secondary Outcome: Change in Total Cholesterol
Description: Mean change in total cholesterol concentration (mg/dL) from baseline to 12 months
Time Frame: Baseline - 12 Months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO)
Number analyzed (Participants) | 37 | 41
mg/dL | 4.22 (12.18) | -8.59 (31.95)
Statistical Analysis 1: Comparison: Basic Resources and Services vs Coordinated Primary Care Population Management (C3PO); Test type: Superiority; p = .02, t-test, 2 sided

6. Secondary Outcome: Change in Non-HDL Cholesterol
Description: Mean change in non-HDL cholesterol concentration (mg/dL) from baseline to 12 months
Time Frame: Baseline - 12 Months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO)
Number analyzed (Participants) | 37 | 41
mg/dL | 4.14 (13.80) | -9.54 (29.92)
Statistical Analysis 1: Comparison: Basic Resources and Services vs Coordinated Primary Care Population Management (C3PO); Test type: Superiority; p = .01, t-test, 2 sided

7. Secondary Outcome: Body Mass Change at 6 Months
Description: Mean Change in Body Mass (kg) from Baseline to 6 Months
Time Frame: Baseline - 6 Months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO)
Number analyzed (Participants) | 36 | 41
kg | -4.19 (7.89) | -1.22 (9.15)
Statistical Analysis 1: Comparison: Basic Resources and Services vs Coordinated Primary Care Population Management (C3PO); Test type: Superiority; p = .13, t-test, 2 sided

8. Secondary Outcome: Body Mass Change at 12 Months
Description: Mean Change in Body Mass (kg) from Baseline to 12 Months
Time Frame: Baseline - 12 Months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO)
Number analyzed (Participants) | 36 | 41
kg | -3.16 (11.66) | -1.87 (10.99)
Statistical Analysis 1: Comparison: Basic Resources and Services vs Coordinated Primary Care Population Management (C3PO); Test type: Superiority; p = .61, t-test, 2 sided

9. Secondary Outcome: Number of Participants Who Achieved 5% Weight Loss Goal in 12 Months
Description: Proportion of Participants who Reach a 5% Weight Loss Goal at 12 Months, calculated as the percent of all participants for whom the following calculation is greater than or equal to 5%: (Baseline body mass (kg) - Body mass measured at 12 months (kg))/(Baseline body mass (kg))
Time Frame: Baseline - 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO)
Number analyzed (Participants) | 38 | 42
Participants | 7 | 10
Statistical Analysis 1: Comparison: Basic Resources and Services vs Coordinated Primary Care Population Management (C3PO); Test type: Superiority; p = .56, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 year following trial enrollment.
Groups:
- Coordinated Primary Care Population Management (C3PO): Patients received outreach engagement in goal setting via MyChart, an electronic scale, telemonitoring of self weighing, information about linkages to extant intensive lifestyle interventions, and outreach MyChart messages that are tailored to each individual's pattern of self-weighing and progress towards their weight goal, and more intensive support from a primary care nurse based on self-weighing behavior and weight loss success.
  .
Arm/Group | Basic Resources and Services | Coordinated Primary Care Population Management (C3PO)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/42
Other Adverse Events (participants affected / at risk) | 0/38 | 0/42

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic began 6-10 weeks into the 12-week active intervention phase. The Illinois stay-at-home order interfered with access to intervention resources as fitness facilities were closed for several months. It also interfered with completion of healthcare visits where follow-up weight measures are captured. Outcome effects observed in this context may not be generalizable if replicated after the Coronavirus pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT03998046/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT03998046/SAP_001.pdf